CLINICAL TRIAL: NCT01279668
Title: A Double Blind Randomised Placebo Controlled Trial of Montelukast in the Treatment of Acute Persistent Cough in Young People and Adults in Primary Care
Brief Title: Montelukast for Persistent Cough in Young People and Adults
Acronym: MAC
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Oxford (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MAC_001; 2010-019647-19 (EudraCT Number)
Record Dates: First submitted 2011-01-17; First posted 2011-01-19 (Estimated); Last update posted 2012-10-10 (Estimated); Status verified 2012-10

CONDITIONS: Persistent Cough; Whooping Cough
Keywords: Montelukast; Persistent cough; Adults; Double-blind randomised placebo controlled trial
MeSH Terms: conditions — Chronic Cough; Whooping Cough | interventions — montelukast

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Montelukast (Experimental)
  Interventions: Drug: Montelukast
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Montelukast — 10mg tablets, once per day for 28 days.
  Other Names: Singulair
  Arms: Montelukast
Drug: Placebo — tablets, once per day for 28 days.
  Arms: Placebo

SUMMARY:
Persistent cough is a common symptom, accounting for about 20% of referrals to outpatient chest clinics. Most coughs are caused by self-limiting viral infections such as the common cold. However, 1 in 4 people with a viral infection develop a persistent cough, which can go on for several weeks. Whooping cough is a common cause of persistent cough in young people and adults. Although the whooping cough vaccine gives lifelong protection against severe infection, it does not appear to give such long-term protection against milder infections, which can make someone cough for many weeks. There are currently no proven efficacious treatments for persistent cough following either a viral infection or infection with whooping cough.

Montelukast is a medication which is already licensed for the treatment of asthma. It works by blocking the action of chemicals called leukotrienes, which make the airways of people with asthma inflamed and sensitive. There is strong evidence to suggest that leukotrienes are also involved in causing persistent cough following viral or whooping cough infection. Montelukast may therefore also help settle persistent coughs in these settings.

Over 18 months, we will recruit patients aged 16-49 years with a cough lasting 2-8 weeks from general practices in England. An oral fluid sample will be taken from each participant to be tested for whooping cough. Participants will be randomly allocated to receive a 28-day course of montelukast or placebo tablets and asked to complete a daily cough diary for two weeks. They will be assessed after two weeks by their GP (face-to-face) and after four weeks by another member of practice clinical staff (telephone). Some participants will be given a 24-hour cough monitor to wear on study entry and at two-week follow-up. This study will be funded by the National Institute for Health Research's School of Primary Care.

ELIGIBILITY:
Inclusion Criteria:

* Male or Female, aged 16 years to 49 years inclusive.
* Presenting with a persistent cough of 2-8 weeks' duration without an established diagnosis (e.g. asthma, gastro-oesophageal reflux).
* Able to complete cough diary and study questionnaires.

Exclusion Criteria:

* There is a contraindication to montelukast.
* Chronic severe disease which may cause persistent cough (eg cystic fibrosis, bronchiectasis, cardiac failure).
* Immunodeficiency/immunocompromised state.
* Pregnancy.
* Breastfeeding.
* Current smoker (i.e. stopped smoking less than 6 months ago).
* Regular medication associated with persistent cough (ACE inhibitors).
* The individual is in another clinical research study.

Ages: 16 Years to 49 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 276 (Actual)
Dates: Start 2011-05; Primary Completion 2012-10 (Estimated); Study Completion 2012-11 (Estimated)

PRIMARY OUTCOMES:
Change in Leicester Cough Questionnaire (LCQ) total score at 2 and 4 weeks post randomisation. | 2 and 4 weeks post randomisation

SECONDARY OUTCOMES:
Change in Leicester Cough Questionnaire (LCQ) physical, psychological and social domain scores at 2 and 4 weeks post randomisation. | 2 and 4 weeks post randomisation
Overall cough severity according to cough visual analogue scale (VAS) scores over the 2-week period post randomisation (area under the curve). | 2 weeks post randomisation
Paroxysmal cough severity over the 2-week period post randomisation (area under the curve). | 2 weeks post randomisation
Proportions of participants reporting cessation of cough at 2 and 4 weeks post randomisation. | 2 and 4 weeks post randomisation
Recruitment rate among young people and adults presenting with acute persistent cough. | End of study
Follow-up rates at 2 weeks and 4 weeks post randomisation. | 2 weeks and 4 weeks post randomisation.
Medication adherence rates at 2 and 4 weeks post randomisation. | 2 and 4 weeks post randomisation
Prevalence of whooping cough among participants. | End of study
Correlations between subjective cough outcome measures (diary-recorded paroxysms of cough, cough visual analogue scale score and exercise-related cough score) and objective cough frequency measured using the Leicester Cough Monitor. | 2 and 4 weeks post randomisation
Proportions of participants undergoing further intervention (re-consultation, investigation, prescription of other medication). | 4 - 8 weeks
  Patient notes will be reviewed in this time frame
Proportions of participants with adverse events. | End of study

CONTACTS AND LOCATIONS:
Overall Officials: Anthony R Harnden, Principal Investigator — University of Oxford
Locations (1):
- University of Oxford, Oxford, Oxfordshire, United Kingdom

REFERENCES:
- [Background] Harnden A, Grant C, Harrison T, Perera R, Brueggemann AB, Mayon-White R, Mant D. Whooping cough in school age children with persistent cough: prospective cohort study in primary care. BMJ. 2006 Jul 22;333(7560):174-7. doi: 10.1136/bmj.38870.655405.AE. Epub 2006 Jul 7. PMID 16829538
- [Background] Birring SS, Prudon B, Carr AJ, Singh SJ, Morgan MD, Pavord ID. Development of a symptom specific health status measure for patients with chronic cough: Leicester Cough Questionnaire (LCQ). Thorax. 2003 Apr;58(4):339-43. doi: 10.1136/thorax.58.4.339. PMID 12668799
- [Derived] Wang K, Birring SS, Taylor K, Fry NK, Hay AD, Moore M, Jin J, Perera R, Farmer A, Little P, Harrison TG, Mant D, Harnden A. Montelukast for postinfectious cough in adults: a double-blind randomised placebo-controlled trial. Lancet Respir Med. 2014 Jan;2(1):35-43. doi: 10.1016/S2213-2600(13)70245-5. Epub 2013 Dec 2. PMID 24461900